CLINICAL TRIAL: NCT03257553
Title: Role of Ultrasound ,Doppler and Calprotectin in Diagnosis of Necrotizing Enterocolitis in Neonates
Brief Title: Ultrasound, Doppler ,and Calprotectin in Necrotizing Enterocolitis Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azhar Arabi mohammed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UDFNEC
Record Dates: First submitted 2017-08-14; First posted 2017-08-22 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Echocardiography, Doppler; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): do fecal calprotectin, doppler and ultrasound for each patient
  Interventions: Diagnostic Test: fecal calprotectin , doppler and ultrasound

INTERVENTIONS:
Diagnostic Test: fecal calprotectin , doppler and ultrasound — faecal sample for measurement of calprotectin level ultrasound and doppler

SUMMARY:
Necrotizing enterocolitis continues to be a disease that is associated with significant morbidity and mortality in premature infants due to advances in neonatal intensive care that increase the survival rate of extremely low birth weight infants (below 1,000 gram)

DETAILED DESCRIPTION:
Necrotizing enterocolitis continues to be a disease that is associated with significant morbidity and mortality in premature infants. It affects annually 0.72 infants per 1000 live births among all neonates and 33 infants per 1000 live births among very low-birth-weight (below 1500 gram).

Necrotising enterocolitis presents with both gastrointestinal and systemic signs. Gastrointestinal signs as delayed gastric emptying, abdominal distention and bloody stools. Non specific signs as lethargy, apnea, respiratory distress.

Although clinical and characteristic radiological findings remain the most important tools so far. Unfortunately, these signs are usually detectable in an advanced stage of disease.

* Haematological studies as severe or persistent thrombocytopenia, neutropenia, coagulopathy, or acidosis might indicate severe disease.
* Serial C-reactive protein : that persistently high C-reactive protein indicated developing complications, such as stricture or abscess.

Unfortunately, the majority of these biomarkers lack accuracy in preclinical stage and do not allow proper discrimination from sepsis Therefore, the search for disease-specific, early and noninvasive diagnostic biomarkers remains warranted.

Calprotectin, a peptide secreted by neutrophils and macrophages and is a useful laboratory biomarker for diagnosing necrotizing enterocolitis . Its non-specific biomarkers of inflammation, but the nature of the specimen, e.g. stool, renders these mediators more indicative of the site of tissue injury. And its levels may be a marker for early diagnosis and resolution of gastrointestinal illness , but its utility for early diagnosis and assessment of resolution of necrotizing enterocolitis needs to be studied in a larger studies.

Plain X ray: Definite signs include pneumatosis intestinalis (intramural air) and portal venous gas .

Ultrasound : More sensitive and accurate imaging studies and could become helpful adjuncts to abdominal films in the diagnosis of necrotizing enterocolitis .

The major advantage of sonography over plain abdominal radiography is its superiority in depicting small amount of gas. Ultrasound with Doppler might be more sensitive than abdominal films for detecting necrotic bowel requiring surgical intervention.

When necrotizing enterocolitis is suspected, infants are given bowel rest , bowel decompression, and broad-spectrum antibiotics (after cultures are obtained). Anaerobic coverage should be considered. Adjunctive therapy includes cardiovascular, pulmonary, and haematological support as clinically indicated.

The two main options available for the surgical management of necrotizing enterocolitis are exploratory laparotomy and primary peritoneal drainage .

ELIGIBILITY:
Inclusion Criteria:

* Include All cases with necrotizing enterocolitis (NEC) in assiut university neonatal intensive care unit (NICU) who are presented with any stage of Bell's stages of necrotising enterocolitis within one year .

I. Suspected disease Mild systemic signs (apnoea, bradycardia, temperature instability) Mild intestinal signs (abdominal distention, gastric residuals, bloody stools) Non-specific or normal radiological signs II. Definite disease Mild to moderate systemic signs Additional intestinal signs (absent bowel sounds, abdominal tenderness) Specific radiologic signs (pneumatosis intestinalis or portal venous air) Laboratory changes (metabolic acidosis, thrombocytopaenia) III. Advanced disease Severe systemic illness (hypotension) Additional intestinal signs (striking abdominal distention, peritonitis) Severe radiological signs (pneumoperitoneum) Additional laboratory changes (metabolic and respiratory acidosis, disseminated intravascular coagulopathy).

Exclusion Criteria:surgical problems other than NEC ,NEC beyond neonatal period.

-

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
diagnosis of necrotizing enterocolitis | one year
  diagnosis of necrotizing enterocolitis by ultrasound, doppler and calprotectin and compare to see more sensitive and specific method of them in comparison with plain erect

CONTACTS AND LOCATIONS:
Overall Officials: Azhar Arabi, MD, Principal Investigator — Assiut University